CLINICAL TRIAL: NCT05706896
Title: Atrophic Age-related Macular Degeneration (AMD) Treated With Intravitreal Injections of Umbilical Cord Blood Platelet-rich Plasma (CB-PRP): a Pilot Study
Brief Title: Atrophic Age-related Macular Degeneration Treated With Intravitreal Injections of Umbilical Cord Blood Platelet-rich Plasma
Acronym: CORD-IV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4995
Record Dates: First submitted 2023-01-09; First posted 2023-01-31 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Dry Age-related Macular Degeneration

STUDY DESIGN:
Intervention Model Description: Randomization will take place by eye, each patient will have one eye treated and the contralateral subjected to sham. The treated eye will receive CB-PRP injections modulated differently over time in each of the sub-studies, i.e. monthly, bimonthly or quarterly, while the contralateral eye will receive a SHAM injection.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Monthly injection (Experimental): The patients will recive 12 intravitreal injections in one eye and 12 sham injections in the other eye each month
  Interventions: Procedure: Intravitreal injection of CB-PRP
- Bimonthly injection (Experimental): The patients will receive 6 intravitreal injections in one eye and 6 sham injections in the other eye each two months
  Interventions: Procedure: Intravitreal injection of CB-PRP
- Quarterly injection (Experimental): The patients will receive 4 intravitreal injections in one eye and 4 sham injections in the other eye each three months
  Interventions: Procedure: Intravitreal injection of CB-PRP

INTERVENTIONS:
Procedure: Intravitreal injection of CB-PRP — The procedure consists in a trans-scleral puncture to access the vitreous cavity, with subsequent injection of CB-PRP
  Other Names: CB-PRP

SUMMARY:
The objective of the study will be to evaluate the efficacy of intravitreal injections of Umbilical Cord Blood Platelet-rich Plasma (CB-PRP) in order to reduce or stabilize the atrophic progression in dry Age-related Macular Degeneration (AMD)

ELIGIBILITY:
Inclusion Criteria:

* Age ≥65 years
* Bilateral dry-AMD
* ETDRS-corrected visual acuity between (or equal to) 1/10 and 4/10
* No concomitant ocular pathology (e.g., Glaucoma, amblyopia) or systemic pathology that would result in a BIAS for primary goal assessment
* Signature of informed consent

Exclusion Criteria:

* Age < 65 years
* Pregnancy
* Previous inflammatory/infectious events involving the eyes
* Eye trauma, diabetes, or disease potentially damaging to the visual system, even in the absence of impairment at the time of intake
* Previous intravitreal treatments.
* Refusal to sign informed consent.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-12-14 (Actual); Primary Completion 2023-06-09 (Actual); Study Completion 2026-02-10 (Estimated)

PRIMARY OUTCOMES:
Autofluorescence atrophy area changes in treated eyes compared with sham group | 1 year
  Stabilization of enlargement of hypoautofluorescent area (atrophy) or at most a maximum increase of no more than 20% compared with baseline in treated subjects compared with placebo group from baseline until follow-ups
Autofluorescence atrophy area changes in treated eyes compared with sham group (1) | 1 year
  Stabilization of the enlargement of the hyperfluorescent area (atrophy enhancement) or at most a maximum increase of not more than 20% from the baseline

SECONDARY OUTCOMES:
ETDRS visual acuity | 1 year
  Increase of at least two lines from baseline measurement and/or to the contralateral untreated eye at 3 and 6, 12, months.
Mean increase in ONL thickness and retinal volumetrics | 1 year
  Mean increase, measured by high-resolution quantitative OCT, of at least 20% from baseline at 3 and 6, 12, months
Mean increase in retinal volumetrics | 1 year
  Mean increase, measured by high-resolution quantitative OCT, of at least 20% from baseline at 3 and 6, 12, months
Stabilization of the atrophy region of the EPR | 1 year
  Stabilization in enface OCT with less than 20% increase from baseline, comparing it with the placebo group, at 3 and 6, 12, months.
Retinography of the ocular fundus | 1 year
  Change in ocular fundus
Incomplete retinal pigment epithelial (RPE) and outer retinal atrophy (iRORA) | 1 year
  Change during follow ups
Outer retinal atrophy (iRORA) | 1 year
  Change during follow ups

OTHER OUTCOMES:
Evaluation of therapy safety | 1 year
  Evaluation of major ocular adverse events (bacterial or fungal septic endophthalmitis, retinal detachment, vitreous proliferative-fibrotic reaction with retinal traction, secondary glaucoma, phthisis bulbs, iris rubeosis), studied at slit-lamp evaluation in the anterior and posterior chambers.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Cristina savastano, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome, Italy

IPD SHARING:
Plan to Share IPD: No